CLINICAL TRIAL: NCT02569658
Title: Investigation of the Blood Sparing Properties of Intravenous Tranexamic Acid With Anatomic and Reverse Total Shoulder Arthroplasty
Brief Title: Investigation of Intravenous Tranexamic Acid With Anatomic and Reverse Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rush TXA TSA
Record Dates: First submitted 2015-10-03; First posted 2015-10-07 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Blood Loss; Anatomic Total Shoulder Arthroplasty; Reverse Total Shoulder Arthroplasty; Transfusion; Tranexamic Acid
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid Group (Experimental): Group will be administered 1 gram tranexamic acid IV bolus (10 ml solution) 10 minutes prior to incision.
  Interventions: Drug: Tranexamic Acid
- Placebo Group (Placebo Comparator): Group will be administered 10 ml normal saline placebo IV bolus 10 minutes prior to incision
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid Group
Drug: Placebo
  Arms: Placebo Group

SUMMARY:
To compare intravenous Tranexamic Acid (TXA) versus normal saline placebo to determine whether or not TXA administration reduces blood loss, decrease in hemoglobin, and rate of transfusions following anatomic and reverse total shoulder arthroplasty (TSA) surgeries.

DETAILED DESCRIPTION:
Anatomic and reverse total shoulder arthroplasty (TSA) is associated with the risk of moderate to significant blood loss that can lead to transfusions. Average estimated blood loss has been reported in the range of 354 to 361 mL intraoperatively, not accounting for additional postoperative blood loss postoperatively in surgical drains. Transfusion rates have been reported to range from 2.4% to 9.5% in recent studies, with rates over 30% for revision cases. Tranexamic acid (TXA) is a synthetic antifibrinolytic agent that is an established method of reducing blood loss and transfusion requirement for patients undergoing total hip and knee arthroplasty. TXA can be administered intravenously, topically (intraarticularly), or orally, with most available literature addressing intravenous and topical administration. Systematic reviews and meta-analyses of the total hip and knee arthroplasty literature demonstrate approximately a 30% decrease in blood loss and 50% decrease in transfusion rate with topical or intravenous administration of TXA compared to placebo. Moreover, the literature demonstrates no increased rate of thromboembolic or other complications associated with TXA administration for hip and knee arthroplasty.

Despite proven efficacy in the hip and knee arthroplasty literature, there have been no studies analyzing the ability of TXA to reduce blood loss and transfusion rate following TSA.

Purpose of the study is to compare intravenous Tranexamic Acid (TXA) versus normal saline placebo to determine whether or not TXA administration reduces blood loss, decrease in hemoglobin, and rate of transfusions following anatomic and reverse total shoulder arthroplasty (TSA) surgeries. With the hypothesis that intravenous TXA will reduce blood loss following TSA.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled for a primary anatomic or reverse TSA

Exclusion Criteria:

* Allergy to TXA
* Acquired disturbances of color vision
* Pre-op use of anticoagulant therapy within five days before surgery
* History of arterial or venous thromboembolic disease; such as DVT, PE, CVA, TIA
* Pregnancy or breastfeeding
* Recent MI (within 6 months of surgery) or any placement of stent regardless of time since placement
* Renal impairment
* Refusal of blood products
* Any patient undergoing a revision TSA
* Patients who decline to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cvetanovich, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Saltzman BM, Chalmers PN, Gupta AK, Romeo AA, Nicholson GP. Complication rates comparing primary with revision reverse total shoulder arthroplasty. J Shoulder Elbow Surg. 2014 Nov;23(11):1647-54. doi: 10.1016/j.jse.2014.04.015. Epub 2014 Jun 28. PMID 24986694
- [Background] Chalmers PN, Gupta AK, Rahman Z, Bruce B, Romeo AA, Nicholson GP. Predictors of early complications of total shoulder arthroplasty. J Arthroplasty. 2014 Apr;29(4):856-60. doi: 10.1016/j.arth.2013.07.002. Epub 2013 Aug 6. PMID 23927910
- [Background] Gupta AK, Chalmers PN, Rahman Z, Bruce B, Harris JD, McCormick F, Abrams GD, Nicholson GP. Reverse total shoulder arthroplasty in patients of varying body mass index. J Shoulder Elbow Surg. 2014 Jan;23(1):35-42. doi: 10.1016/j.jse.2013.07.043. Epub 2013 Sep 30. PMID 24090984
- [Background] Shields E, Iannuzzi JC, Thorsness R, Noyes K, Voloshin I. Perioperative complications after hemiarthroplasty and total shoulder arthroplasty are equivalent. J Shoulder Elbow Surg. 2014 Oct;23(10):1449-53. doi: 10.1016/j.jse.2014.01.052. Epub 2014 Apr 18. PMID 24751531
- [Background] Yang ZG, Chen WP, Wu LD. Effectiveness and safety of tranexamic acid in reducing blood loss in total knee arthroplasty: a meta-analysis. J Bone Joint Surg Am. 2012 Jul 3;94(13):1153-9. doi: 10.2106/JBJS.K.00873. PMID 22623147
- [Background] Gandhi R, Evans HM, Mahomed SR, Mahomed NN. Tranexamic acid and the reduction of blood loss in total knee and hip arthroplasty: a meta-analysis. BMC Res Notes. 2013 May 7;6:184. doi: 10.1186/1756-0500-6-184. PMID 23651507
- [Background] Alshryda S, Mason J, Sarda P, Nargol A, Cooke N, Ahmad H, Tang S, Logishetty R, Vaghela M, McPartlin L, Hungin AP. Topical (intra-articular) tranexamic acid reduces blood loss and transfusion rates following total hip replacement: a randomized controlled trial (TRANX-H). J Bone Joint Surg Am. 2013 Nov 6;95(21):1969-74. doi: 10.2106/JBJS.L.00908. PMID 24196467
- [Background] Alshryda S, Mason J, Vaghela M, Sarda P, Nargol A, Maheswaran S, Tulloch C, Anand S, Logishetty R, Stothart B, Hungin AP. Topical (intra-articular) tranexamic acid reduces blood loss and transfusion rates following total knee replacement: a randomized controlled trial (TRANX-K). J Bone Joint Surg Am. 2013 Nov 6;95(21):1961-8. doi: 10.2106/JBJS.L.00907. PMID 24196466
- [Background] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid Group: Group will be administered 1 gram tranexamic acid IV bolus (10 ml solution) 10 minutes prior to incision.
  Tranexamic Acid
- Placebo Group: Group will be administered 10 ml normal saline placebo IV bolus 10 minutes prior to incision
  Placebo
Period: Overall Study
Arm/Group | Tranexamic Acid Group | Placebo Group
Started | 53 | 57
Completed | 52 | 56
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Group | Placebo Group | Total
Number analyzed (Participants) | 52 | 56 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (10.9) | 65.2 (9.2) | 66.4 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 23 | 28 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: kg] | 84.2 (19.6) | 88.4 (19.1) | 86.4 (19.3)
operative time [Mean (Standard Deviation); unit: minutes] | 101.1 (21.4) | 102.7 (21.6) | 101.9 (21.5)
reverse total shoulder arthroplasty [Count of Participants; unit: Participants] | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Blood Loss
Description: Equated based on the patient's predicted blood volume and change in hemoglobin from the pre-operative level to the lowest post-operative level.
Time Frame: Average of 3 days post-operatively
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 52 | 56
mL | 152.2 (57.3) | 178.0 (65.8)

2. Secondary Outcome: Number of Units Transfused
Description: Units of pack red blood cells that the patients recieved
Time Frame: Average of 3 days post-operatively
Measure: Number; unit: Units of PRBCs
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 52 | 56
Units of PRBCs | 0 | 0

3. Secondary Outcome: Number of Patients Transfused
Description: Patients who received a post-op transfusion of pack red blood cells
Time Frame: Average of 3 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 52 | 56
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Deep Vein Thrombosis
Description: Must be diagnosed via ultrasound duplex
Time Frame: 30 days post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 52 | 56
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With Pulmonary Embolism
Description: Must be diagnosed via CT chest or V/Q lung scan
Time Frame: 30 days post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 52 | 56
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Stroke
Description: Must be diagnosed via CT scan or MRI
Time Frame: 30 days post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Group | Placebo Group
Number analyzed (Participants) | 52 | 56
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days post-operative
Arm/Group | Tranexamic Acid Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/56
Other Adverse Events (participants affected / at risk) | 0/52 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid Group (N=52) | Placebo Group (N=56)
DVT (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT02569658/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT02569658/ICF_001.pdf